CLINICAL TRIAL: NCT07049484
Title: Clinical and Biomechanical Outcomes of Anterior Cruciate Ligament (ACL) Reconstruction Associated With Lateral Extra-articular Tenodesis (LET): a Short-term Prospective Arthrometric Study
Brief Title: Clinical and Biomechanical Outcomes of Anterior Cruciate Ligament (ACL) Reconstruction Associated With Lateral Extra-articular Tenodesis (LET)
Acronym: LETOTT
Status: Not yet recruiting | Type: Observational
Sponsor: Stefano Zaffagnini (Other)
Responsible Party: Sponsor-Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: LETOTT
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: ACL Reconstruction; Tenodesis; ACL Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The anterior cruciate ligament (ACL) is one of the main stabilizers of the knee joint, and its injury is among the most common soft tissue injuries of the knee. Several surgical reconstruction techniques are available, utilizing various tissues as a graft for the neo-ligament, including both autografts and allografts.

The "Over-the-top single-bundle technique with gracilis and semitendinosus tendons combined with lateral extra-articular tenodesis (LET)" was developed in 1998 by Prof. Marcacci and Prof. Zaffagnini, and it is still the preferred method for ACL reconstruction at the Second Clinic of the Rizzoli Orthopaedic Institute.

Cadaveric biomechanical studies have shown that combining LET with ACL reconstruction improves knee joint stability in both the anteroposterior and rotational planes. However, a recent in vivo study has challenged this hypothesis, showing that in patients undergoing surgery, the addition of LET enhances knee stability only in the anteroposterior direction and only for a limited period of six months. At twelve months postoperatively, joint laxity appeared similar to that of patients who did not undergo the additional procedure. Furthermore, the same study did not assess rotational instability using the pivot-shift test, an essential parameter as it is closely linked to knee stability and the patient's subjective perception of surgical success.

Despite the increasing use of LET in conjunction with ACL reconstruction, few studies have analyzed the short-term postoperative effects of lateral extra-articular tenodesis and its potential benefits during the early stages of rehabilitation and return to sport.

This study was conceived in response to this clinical question, with the goal of evaluating anteroposterior and rotational laxity in a group of patients who underwent ACL reconstruction combined with LET, in order to analyze clinical outcomes and, most importantly, any changes in stability during the early postoperative period.

The results aim to improve understanding of knee stability in the initial phase following surgery, providing valuable information for rehabilitation teams to optimize recovery protocols and more effectively guide return-to-sport decisions for patients undergoing both procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isolated ACL reconstruction using gracilis and semitendinosus tendons with the over-the-top technique and LET.
* Both male and female patients.
* Patients who have given consent to participate in the study.
* Age between 18 and 50 years at the time of surgery.

Exclusion Criteria:

* Previous surgery on the same limb (meniscectomy, prior ACL reconstruction, displaced fractures).
* Surgical technique different from Over-the-Top with LET using autologous gracilis and semitendinosus tendons.
* Other concomitant ligament injuries requiring surgical treatment.
* Patients undergoing additional procedures at the same time as ACL reconstruction and LET (e.g., concomitant osteotomy, meniscus transplant, cartilage procedure…).
* Patients who did not provide informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be recruited from those surgically treated at the Second Clinic of the Rizzoli Orthopaedic Institute, undergoing anterior cruciate ligament reconstruction using the "over-the-top" single-bundle technique with gracilis and semitendinosus tendons, combined with lateral extra-articular tenodesis (LET). Only patients with at least 6 months of follow-up after the surgery date will be enrolled. Subsequently, patients will be re-evaluated during a 12-month follow-up visit, as per standard clinical practice for this procedure.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
KYRA accelerometer | 12 months
  KYRA is a non-invasive outpatient device that allows the assessment of dynamic laxity during the pivot shift phenomenon. The device enables highly precise quantification of the degree of laxity. The unit of measurement is millimeters per second squared.

SECONDARY OUTCOMES:
KT-1000 Arthrometer | 12 months
  The KT-1000 is an objective assessment tool that measures anterior tibial translation relative to the position of the femur by applying a predefined force that pushes the tibia forward. It is commonly used in research settings to quantitatively evaluate static anteroposterior knee laxity following anterior cruciate ligament reconstruction surgeries.
Physical Examination | 12 months
  A standard physical examination will be performed, including palpation, assessment of joint mobility, and laxity. During palpation, the typical tender points related to meniscal pathology are examined: the joint line areas on their anterior, middle, and posterior aspects. Pain is recorded as either present or absent. Joint mobility is assessed by asking the patient to flex and extend the knee, measuring the angle formed in degrees (0-130), with attention to the presence or absence of any joint clicks or catches. Laxity is evaluated using the classic tests: anterior drawer test, Lachman test, and pivot shift test.
Anterior Drawer Test | 12 months
  This test allows evaluation of the anterior translation of the tibia relative to the femur with the knee flexed at 90 degrees. An increased translation suggests a lesion of the reconstructed ACL (neo-ACL). The degree of translation is quantified on a scale from 0 to 3.
Lachman Test | 12 months
  This test allows evaluation of the anterior translation of the tibia relative to the femur with the knee flexed at 30 degrees. An increased translation suggests a lesion of the reconstructed ACL (neo-ACL). It is quantified on a scale from 0 to 3.
Pivot Shift Test | 12 months
  This is a clinical maneuver used to assess rotational instability of the knee under examination. The test is performed by applying an internal rotation, valgus stress, and knee flexion; the occurrence of a tibial "clunk" or shift suggests a lesion of the reconstructed ACL (neo-ACL) associated with rotational instability. It is quantified on a scale from 0 to 3.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 12 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a self-administered questionnaire used to evaluate both short- and long-term outcomes after a knee injury. It assesses five dimensions: pain, symptoms, activities of daily living, sports and recreational function, and knee-related quality of life.
  Each dimension is scored separately using a 5-point Likert scale ranging from 0 (no problems) to 4 (extreme problems). Scores for each dimension are summed and then transformed to a 0-100 scale, where 0 represents extreme knee problems and 100 indicates no knee problems. The KOOS meets essential standards for outcome measures and is useful for monitoring the progression of knee injuries and the effectiveness of treatments.
Lysholm Knee Score | 12 months
  The Lysholm Knee Score is a validated measurement scale that evaluates knee function through 8 items, allowing assessment of the knee's condition in relation to the functional demands of daily activities. This assessment tool is used to evaluate surgical outcomes in patients operated on for ligament or meniscal injuries of the knee. The final score is obtained by summing the scores from the different items and ranges from 0 to 100. Scores are categorized into subgroups: Excellent (95-100), Good (84-94), Fair (65-83), and Poor (<64).
VAS (Visual Analog Scale) | 12 months
  The VAS is a unidimensional quantitative numerical scale for pain assessment ranging from 0 to 10. The patient selects the number that best describes the intensity of their pain at that moment. A score of 0 means no pain, and 10 indicates the worst possible pain.
Tegner Score | 12 months
  The Tegner Score estimates a person's level of physical activity on a scale from 0 to 10, where 0 represents "disability" and 10 represents participation in competitive sports, such as national or international-level soccer. This score is the most widely used to define the physical activity level of patients with knee disorders. In the study, the Tegner Score will be completed directly by the examiner through an interview with the patient.
Complications or Subsequent Interventions | 12 months
  Any complications and subsequent interventions will be documented and recorded in the Case Report Form (CRF). The staff responsible for distributing and collecting the questionnaires will assign an identification code on the questionnaire cover page to protect the privacy of the study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy